CLINICAL TRIAL: NCT01716598
Title: IPS-II Study: Evaluation of the Innovative Pulmonary Solutions (IPS) System for Targeted Lung Denervation (TLD) Therapy in Patients With Chronic Obstructive Pulmonary Disease (COPD) - A Pilot Study.
Brief Title: Evaluation of the IPS System for TLD Therapy in Patients With COPD
Acronym: IPS-II
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nuvaira, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-002; CVI-12-03-005102 (Other: Eudamed Number)
Record Dates: First submitted 2012-10-04; First posted 2012-10-30 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; TLD Therapy; Targeted Lung Denervation Therapy; IPS; Innovative Pulmonary Solutions, Inc.; Holaira, Inc.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Targeted Lung Denervation Therapy (TLD Therapy)
  Interventions: Device: IPS System

INTERVENTIONS:
Device: IPS System — TLD Therapy will be achieved bronchoscopically.
  Other Names: TLD Therapy; Targeted Lung Denervation Therapy

SUMMARY:
Targeted Lung Denervation (TLD) Therapy will be a safe method to ablate the airway nerve trunks that travel parallel to and outside of the main bronchi and into the lungs to achieve targeted lung denervation and potentially improve breathing and quality of life for patients suffering from COPD.

Use of the IPS System will be technically feasible in accessing the target treatment location and delivering RF energy to the target treatment location.

ELIGIBILITY:
Inclusion Criteria:

* FEV1 30% to 60%
* Patient is diagnosed with COPD
* Positive relative change in FEV1 of greater than 15%
* Patient 40 years of age or older at the time of consent
* Smoking history of at least 10 pack years
* Non-smoking for a minimum of 6 months prior to consent and agrees to continue not smoking for the duration of the study

Exclusion Criteria:

* Documented history or current evidence of pulmonary hypertension Documented history or current evidence of polycythemia level of greater
* Documented history or current evidence of congestive heart failure
* Patient has an SaO2 less than or equal to 88% or a PaO2 less than or equal to 7.3 kPa (55 mm Hg) on room air
* Patient has a PaCO2 > 8.0 kPa (60 mm Hg)
* Prior lung transplant, LVRS, LVR, median sternotomy, bullectomy or lobectomy
* Pulmonary nodule requiring surgery
* History of recurrent respiratory infections (more than 3 hospitalizations within 1 year of enrollment)
* Presence of a pacemaker, internal defibrillator or other implantable electronic devices j. Active respiratory infection within the past 4 weeks k. COPD exacerbation within the past 4 weeks l. Myocardial infarction (MI) within the last 6 months m. Unstable or life threatening arrhythmia within the last year n. Malignancy treated with radiation or chemotherapy within the last 2 years o. Documented history of other respiratory diseases (cystic fibrosis, tuberculosis, vocal chord dysfunction, Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 365 Days
  Safety will be evaluated as freedom from documented and sustained worsening of COPD directly attributable to the investigational device or procedure.

SECONDARY OUTCOMES:
Performance | 365 days
  Performance will be evaluated as the ability of the IPS System to access the target treatment area and deliver RF energy to the target treatment site at the time of the procedure, as well as confirmation of clinical evidence of successful lung denervation.

CONTACTS AND LOCATIONS:
Overall Officials: Arschang Valipour, MD, FCCP, Ass. Prof., Principal Investigator — Otto-Wagner Hospital, Vienna, Austria
Locations (4):
- Otto-Wagner Hospital and Medical Center, Sanatoriumstrasse 2, Vienna, Austria
- France (3):
  - Centre Hospitalier et Universitaire de Grenoble, Grenoble
  - Centre Hospitalier University de Reims, Reims
  - Nouvel Hopital Civil, Strasbourg